CLINICAL TRIAL: NCT00109655
Title: A Phase 1 Dose-Escalation Trial of Intravesical CG0070 for Superficial Transitional Cell Carcinoma of the Bladder After Bacillus Calmette-Guerin Failure
Brief Title: Dose-Escalation Study of CG0070 for Bladder Cancer After BCG (Bacillus Calmette-Guerin) Failure
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cell Genesys (Industry)
Responsible Party: Cell Genesys, Inc, Cell Genesys, Inc
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V-0046
Record Dates: First submitted 2005-05-02; First posted 2005-05-03 (Estimated); Last update posted 2008-10-03 (Estimated); Status verified 2008-10

CONDITIONS: Carcinoma, Transitional Cell; Bladder Neoplasms
Keywords: Superficial Transitional Cell Carcinoma; Bacillus Calmette-Guerin (BCG); Superficial Bladder Cancer; Gene Therapy; Vaccine; Adenovirus; Carcinoma in situ
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Adenoviridae Infections; Carcinoma in Situ

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Oncolytic adenovirus (serotype 5) - CG0070

INTERVENTIONS:
Biological: Oncolytic adenovirus (serotype 5) - CG0070 — Intravesical administration of CG0070 (in suspension) directly into the bladder

SUMMARY:
The main purpose of this research study is to evaluate the safety and dosing of CG0070.

DETAILED DESCRIPTION:
Cohorts of three to six patients will be assigned to receive intravesical (into the bladder) administration of CG0070 either Weekly or Every 4 Weeks for up to a total of 6 doses.

ELIGIBILITY:
Inclusion Criteria:

* High grade non-muscle invasive bladder cancer (stages Ta, T1 and/or CIS - carcinoma in situ). High grade being defined as G2 or G3 disease.
* Failure of at least one prior treatment with BCG, defined as evidence of TCC on cystoscopic exam and biopsy or cystoscopic exam and urine cytology at least 6 weeks from last BCG treatment
* ECOG performance status 0-1
* Adequate bone marrow, renal, liver and coagulation function

Exclusion Criteria:

* Pregnant or nursing
* HIV positive
* Use of anticoagulants such as coumadin or heparin
* History of bleeding disorder
* Active systemic autoimmune disease or chronic immunodeficiency
* Prior gene therapy
* Uncontrolled cystitis, bladder pain, bladder spasms, urinary incontinence, or reduced bladder volume

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2005-04; Primary Completion 2008-10 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Maximum-tolerated or maximum feasible dose in single and multidose regimens of CG0070 by intravesical administration | Study End

SECONDARY OUTCOMES:
Assessment of the amount of CG0070 in the urine and blood over time by PCR | Study End

CONTACTS AND LOCATIONS:
Locations (10):
- United States (8):
  - BCG Oncology, Phoenix, Arizona
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Billings Clinic, Billings, Montana
  - New York Oncology Hematology, Albany, New York
  - Columbia University, New York, New York
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
- Canada (2):
  - Male/Female Health and Research Centre, Barrie, Ontario
  - The Fe/Male Health Centre, Oakville, Ontario

REFERENCES:
- See also: Related Info — http://www.cellgenesys.com